CLINICAL TRIAL: NCT04883489
Title: Clinical Classification of Musculoskeletal Pain in Caregivers for Children With Cerebral Palsy
Brief Title: Pain Classification in Caregivers for Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Ismail Saracoglu, Principal Investigator, Kutahya Health Sciences University
Other Study IDs: KutahyaHSU pain in caregivers
Record Dates: First submitted 2021-05-07; First posted 2021-05-12 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Chronic Pain; Cerebral Palsy; Musculoskeletal Pain; Caregivers
Keywords: chronic pain
MeSH Terms: conditions — Chronic Pain; Cerebral Palsy; Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The care of children with Cerebral Palsy is a process that continues for many years. Individuals who take care of them experience musculoskeletal pain due to the difficulties they experience and face pain that becomes chronic over time. For individuals who take care of children with CP, determining the types of chronic pain is important in order to clarify the classification criteria and for individuals to reach better living standards by tailoring the treatments they will receive. Therefore, the aim of the study is to determine the types of chronic pain in caregivers for children with cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Having musculoskeletal pain complaints for the last 6 months or more
* experienced musculoskeletal pain or a sensitive disorder (like numbness, tingling, etc.) anywhere in body for which they stated a minimum score of 2 on a numeric pain rating scale
* pain that lasts at least 6 months
* To provide the documented diagnosis of Cerebral palsy of the child in the care of the participants.

Exclusion Criteria:

* Having severe psychological illness
* Having a cognitive dysfunction
* Not participating in the assessment or submitting incomplete answers for questionnaires

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The convenience sampling will implement for this cross-sectional study. Caregivers for children with Cerebral palsy chronic pain who presented at the different Educational and Rehabilitation Center in Kutahya will screen for eligibility by a clinician and will subsequently request to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 1 minute
  The NPRS was used to assess the participants' pain levels. In the NPRS, patients are asked to verbally rate the severity of their pain on a scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Margolis Pain Diagram | 5 minute
  The Margolis Pain Diagram, consists of a dorsal and a ventral drawing body, is used to assess the location and distribution of the pain. Participants will ask to point out the place where they experience pain during the preceding 4 weeks for at least 24 hours
Central Sensitization Inventory | 10 minute
  The Central Sensitization Inventory (CSI) aims to evaluate symptoms thought to be associated with nociplastic pain. The CSI consists 25 items exploring emotional and somatic disorders associated with CS. Each response is scored from 0 to 4, yielding a total score of 0 to 100. A score of 40 or higher on the CSI means the presence of nociplastic pain.
Short Form 36 | 10 minute
  The Short Form-36 (SF-36) is widely used to measurement of health related quality of life (HRQoL) questionnaire. SF-36 is a 36-item generic self-administered instrument consisting of 8 subscales related to various aspects of HRQoL: physical functioning, physical role, bodily pain, general health, vitality, social functioning, emotional role, and mental health. The 8 subscales are scored from 0 to 100, with higher scores indicating better health status.

SECONDARY OUTCOMES:
Quantitative sensory test | 10 minute
  Quantitative sensory testing (QST) is a psychophysical method used to quantify somatosensory function in patients. In QST will be used various stimuli static thermal (thermotest), static mechanical ( a painter brush), pinprick (a calibrated pin) and vibration ( a tuning folk). QST will interrogate whether each stimulus is considered a sensory loss (negative sign) or sensory gain (positive sign or hyperalgesia).

CONTACTS AND LOCATIONS:
Locations (1):
- KutahyaHSU, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided